CLINICAL TRIAL: NCT01765010
Title: Comparisons of the Effect of Inactive and Active Vitamin D on Serum Sclerostin/dickkopf1 Levels
Brief Title: The Effect of Inactive and Active Vitamin D on Serum Sclerostin/dickkopf1 Levels
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SNUH-ENDO-2013
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Osteoporosis
Keywords: Vitamin D; Serum sclerostin; Serum dickkopf1
MeSH Terms: conditions — Osteoporosis | interventions — Calcitriol; Calcium; alfacalcidol; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo control (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo
- Cholecalciferol 1000IU (Active Comparator): Cholecalciferol 1000IU qd for 8 weeks
  Interventions: Drug: Cholecalciferol
- alfacalcidol (Experimental): alfacalcidol 0.5ug qd for 8 weeks
  Interventions: Drug: Alfacalcidol
- Calcitriol (Experimental): Calcitriol 0.25ug qd for 8 weeks
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Calcitriol
  Other Names: Calcio
  Arms: Calcitriol
Drug: Alfacalcidol
  Other Names: Onealfa
  Arms: alfacalcidol
Drug: Cholecalciferol
  Other Names: DicamaxD
  Arms: Cholecalciferol 1000IU
Drug: Placebo
  Arms: Placebo control

SUMMARY:
The purpose of this study is to compare the effect of inactive and active vitamin D on serum sclerostin and dickkopf1 levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteer older than 20 years

Exclusion Criteria:

* Subjects with bone and mineral metabolism disorders
* Subjects with kidney or liver diseases
* Subjects with uncorrectable hypercalcemia or hypocalcemia
* Subjects with chronic gastrointestinal disorders or malabsorption
* Subjects taking medication related to bone loss

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Change of serum sclerostin level | 8 weeks later
Change of serum Dickkopf1 level | 8 weeks later

SECONDARY OUTCOMES:
Change of serum c-telopeptide level | 8 weeks later
Change of serum bone-specific alkaline phosphatase level | 8 weeks later
Change of serum calcium level | 8 weeks later
Change of serum parathyroid hormone level | 8 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Chan Soo Shin, MD, PhD, Principal Investigator — Seoul National University Medical School
Locations (1):
- Seoul National University Medical School, Seoul, South Korea